CLINICAL TRIAL: NCT02745340
Title: Effect of an Acetate-free Dialysis (Citrate Based) on Parameters of Central Hemodynamics, Dialysis Adequacy, Quality of Life and Immunological Parameters in Chronic Hemodialysis
Brief Title: Substitution of Acetate by Citrate in the Bicarbonate Based Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Gambro Renal Products, Inc. (Industry)
Responsible Party: Principal Investigator, PD Dr. Christoph Schmaderer, Study Principal Investigator (Prüfer), Technical University of Munich
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 344/15s
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetate (Active Comparator)
  Interventions: Other: Acetate by Citrate substitution and vice versa
- Citrate (Experimental)
  Interventions: Other: Acetate by Citrate substitution and vice versa

INTERVENTIONS:
Other: Acetate by Citrate substitution and vice versa — substitution of acetate by citrate in dialysis fluid

SUMMARY:
Acetate is the primary acidifying solution used in bicarbonate-based hemodialysis worldwide. It has been published in small trials or case series that the addition of acetate is associated with a rise in nitric oxide production of vascular smooth muscle cells, endothelial cells and myocardial cells as a sign of vascular dysfunction. Furthermore clinical side effects of dialysis e.g. nausea, malnutrition, intradialytic blood pressure drops, induction of proinflammatory cytokines and activation of complement and leukocytes have been described with acetate.

Citrate on the other hand was associated with: Acid-base disorders (metabolic alkalosis), Disturbances of the calcium homeostasis (Hypocalcemia), but also anti-inflammatory effects. Both dialysate additives (citrate and acetate) are commercially available and are used world wide in dialysis centers.

The investigators hypothesize that substitution of acetate by citrate reduces the cardiovascular risk (measured by a change in the surrogate parameter of pulse wave velocity and Augmentation index) and might improves quality of life in the participants. Furthermore the investigators speculate that citrate in the dialysis solution could reduce systemic inflammation in the participants of the study.

ELIGIBILITY:
Inclusion Criteria:

* time since initiation of dialysis > 3 months
* age > 18 years
* dialysis 3x/week for > 4 hrs

Exclusion Criteria:

* ongoing infection
* pregnancy
* lack of written and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in Augmentation Index (AIx) | 6 months (cross over after 3 months)
  cross over design

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schmaderer, M.D., Principal Investigator — attending, board certified nephrologist
Locations (2):
- Germany (2):
  - Nierenzentrum24 NEUPERLACH, Munich, Bavaria
  - Nierenzentrum Bogenhausen, Munich, Bavaria

REFERENCES:
- [Background] Molina Nunez M, de Alarcon R, Roca S, Alvarez G, Ros MS, Jimeno C, Bucalo L, Villegas I, Garcia MA. Citrate versus acetate-based dialysate in on-line haemodiafiltration. A prospective cross-over study. Blood Purif. 2015;39(1-3):181-187. doi: 10.1159/000371569. PMID 25791278